CLINICAL TRIAL: NCT01093495
Title: A Randomized Controlled Trial on Weaning Preterm Neonates From Nasal Continuous Positive Airway Pressure
Brief Title: Weaning Preterm Neonates From Nasal Continuous Positive Airway Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Hesham Abdel Hady, Mansoura University Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20081230
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Respiratory Distress Syndrome; Hyaline Membrane Disease; Preterm Infants; Premature Infants
Keywords: Nasal Continuous positive Airway pressure; Nasal Cannula; CPAP; Premature; RDS; HMD; NICU
MeSH Terms: conditions — Respiratory Distress Syndrome; Hyaline Membrane Disease; Premature Birth | interventions — Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP group (Experimental): Subjects in this group will continue receiving CPAP until no oxygen requirement for 24 hours, then will be weaned off CPAP completely as long as they tolerate. CPAP will be re-instituted if subjects meet failing criteria. Another trial off CPAP will start 24 hours after failure and/or after being on 21% for 24 hours. CPAP will be weaned off directly to room air at all times.
  Interventions: Device: CPAP
- Nasal Cannula Group (Experimental): Subjects will be weaned from CPAP (when FiO2 <0.30) to Nasal cannula (2 L/min) with whatever FiO2 they need until they are off oxygen and NC completely. However, if these infants fail on NC they will be put back to nCPAP. Infants will then be maintained on CPAP until stable on CPAP-30% for 24 hours. Infants will be tried for another weaning using NC. So, infants assigned to NC will be weaned only through NC. CPAP will be used only for stabilization in between trials if needed.
  Interventions: Device: Nasal Cannula

INTERVENTIONS:
Device: CPAP — CPAP
  Arms: CPAP group
Device: Nasal Cannula — Nasal Cannula
  Arms: Nasal Cannula Group

SUMMARY:
There is little data published concerning the best approach to nasal continuous positive airway pressure (nCPAP) weaning. Potential complications associated with prolonged nCPAP therapy include gastric distension, nasal trauma,pneumothorax,agitation and nosocomial infection. Moreover, Infants on nCPAP may also require more intensive nursing care and the use of extra equipment. Therefore, minimizing the amount of time that a patient requires CPAP may be beneficial. On the other hand, removing CPAP too early may lead to complications that include: increasing apnea, increased oxygen requirement, increased work of breathing, the need to re-start CPAP, and intubation and mechanical ventilation. Moreover, an experimental study have demonstrated an improvement in lung growth after the prolonged use of CPAP.

Nasal cannula (NC) flows at 1-2 L/min may also generate a positive pressure in the airway of preterm infants. The use of NC flow to generate positive airway pressure would minimize many of the application issues of nCPAP. However, NC systems used in neonates routinely employ gas that is inadequately warmed and humidified, limiting the use of such flows due to increased risk of nasal mucosa injury, and possibly increasing the risk for nosocomial infection.

The purpose of this randomized controlled trial is to evaluate the clinical impact of two methods for weaning preterm infants from nCPAP.

DETAILED DESCRIPTION:
The objective of this study is to test the null hypothesis that in preterm infants with gestational age of 28 to 36 weeks who are stable on CPAP pressure of 5 cmH2O and with oxygen concentrations (FiO2) <0.30, keeping these infants on CPAP or changing them to NC flow of 1-2 L/min will not make any difference in length of hospitalization, length of respiratory support and incidence of complications.

ELIGIBILITY:
Inclusion Criteria:

* Infants born greater than or equal to 28 weeks (28+0) and less than 37 weeks (36+6) gestation
* CPAP pressure of 5 cm H2O
* FiO2 requirement = or <0.30
* Clinically stable on these CPAP parameters for 24 hours pre-randomization:

  * Respiratory rate less than 60
  * No significant chest recession
  * No apnea requiring bagging and/or
  * Not more than 6 apneas requiring stimulation in the preceding 24 h.
  * Average saturation > or = 87%
  * Satisfactory ABG (pH> 7.25, PCO2 < 60, and Base deficit < -8)

Exclusion Criteria:

* Life threatening congenital anomalies
* Congenital cyanotic heart diseases
* Congenital airway or chest wall abnormalities
* Pulmonary hypoplasia
* Known or suspected to have a neuromuscular disorder
* Congenital neurological disorder, severe IVH (grade 3 or 4), PVL and hydrocephalus

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Duration of oxygen use | 3 months
  The number of days for oxygen use from the start of randomization until hospital discharge will be recorded.

SECONDARY OUTCOMES:
Length of respiratory support | 3 months
  The number of days in which the subject requires any sort of respiratory support will be recorded, including: CPAP, nasal cannula and mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Hesham Abdel Hady, MD, Principal Investigator — Mansoura University Children's Hospital
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Egypt

REFERENCES:
- [Background] Ho JJ, Henderson-Smart DJ, Davis PG. Early versus delayed initiation of continuous distending pressure for respiratory distress syndrome in preterm infants. Cochrane Database Syst Rev. 2002;2002(2):CD002975. doi: 10.1002/14651858.CD002975. PMID 12076463
- [Background] Ho JJ, Subramaniam P, Henderson-Smart DJ, Davis PG. Continuous distending pressure for respiratory distress syndrome in preterm infants. Cochrane Database Syst Rev. 2002;(2):CD002271. doi: 10.1002/14651858.CD002271. PMID 12076445
- [Background] Aly H, Massaro AN, Patel K, El-Mohandes AA. Is it safer to intubate premature infants in the delivery room? Pediatrics. 2005 Jun;115(6):1660-5. doi: 10.1542/peds.2004-2493. PMID 15930230
- [Background] Aly H, Massaro AN, Hammad TA, Narang S, Essers J. Early nasal continuous positive airway pressure and necrotizing enterocolitis in preterm infants. Pediatrics. 2009 Jul;124(1):205-10. doi: 10.1542/peds.2008-2588. PMID 19564301
- [Background] Abdel-Hady H, Matter M, Hammad A, El-Refaay A, Aly H. Hemodynamic changes during weaning from nasal continuous positive airway pressure. Pediatrics. 2008 Nov;122(5):e1086-90. doi: 10.1542/peds.2008-1193. PMID 18977958
- [Background] Aly H. Is there a strategy for preventing bronchopulmonary dysplasia? Absence of evidence is not evidence of absence. Pediatrics. 2007 Apr;119(4):818-20. doi: 10.1542/peds.2006-3026. No abstract available. PMID 17403854
- [Background] Aly H, Massaro AN, El-Mohandes AA. Can delivery room management impact the length of hospital stay in premature infants? J Perinatol. 2006 Oct;26(10):593-6. doi: 10.1038/sj.jp.7211575. Epub 2006 Jul 20. PMID 16855619
- [Background] Aly H, Milner JD, Patel K, El-Mohandes AA. Does the experience with the use of nasal continuous positive airway pressure improve over time in extremely low birth weight infants? Pediatrics. 2004 Sep;114(3):697-702. doi: 10.1542/peds.2003-0572-L. PMID 15342841
- [Derived] Abdel-Hady H, Shouman B, Aly H. Early weaning from CPAP to high flow nasal cannula in preterm infants is associated with prolonged oxygen requirement: a randomized controlled trial. Early Hum Dev. 2011 Mar;87(3):205-8. doi: 10.1016/j.earlhumdev.2010.12.010. Epub 2011 Jan 26. PMID 21276671